CLINICAL TRIAL: NCT00702650
Title: A Phase III Open-label Titration Trial to Evaluate the Effectiveness and Safety of Different Doses of a Dermal Application of Testosterone MD-Lotion® (Cutaneous Solution) in Hypogonadal Men
Brief Title: A Titration Trial to Determine the Effectiveness of Testosterone MD-Lotion (Cutaneous Solution) Formulations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14272; MTE08 (Other: Acrux); I5E-MC-TSAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone MD-Lotion (Experimental): Participants received Testosterone Metered Dose (MD)-Lotion for 120 days. Participants started by receiving 3.0 mL (60 mg) of 2% Testosterone MD-Lotion, and based upon restoration to eugonadal levels, may have had their dose of testosterone adjusted upwards or downwards on Days 45 and 90.
  Doses could be titrated to one of the following:
  1.5 mL (30 mg) of 2% Testosterone MD-Lotion applied daily by 1 dose to the axilla (1.5 mL to one axilla).
  3.0 mL (60 mg) of 2% Testosterone MD-Lotion applied daily by 2 doses to the axilla (1.5 mL to each axilla).
  4.5 mL (90 mg) of 2% Testosterone MD-Lotion applied daily by 3 doses to the axilla (2 x 1.5 mL to one axilla and 1 x 1.5 mL to the other axilla).
  6.0 mL (120 mg) of 2% Testosterone MD-Lotion applied daily by 4 doses to the axilla (2 x 1.5 mL to each axilla).
  Interventions: Drug: Testosterone MD-Lotion

INTERVENTIONS:
Drug: Testosterone MD-Lotion — 30 mg to 120 mg administered topically once daily for 120 days
  Other Names: LY900011; Axiron

SUMMARY:
Testosterone replacement treatment is the most effective way of treating hypogonadism in men. Acrux has a propriety testosterone replacement product- Testosterone MD-Lotion (cutaneous solution), and this study will evaluate the efficacy via pharmacokinetics of various doses of this product. The study will also assess safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with a prior documented definitive diagnosis of hypogonadism as evidenced by previously documented:

  * Hypothalamic, pituitary or testicular disorder or age related idiopathic hypogonadism
  * Screening serum testosterone of less than or equal to 300 ng/dL (based on the average of two morning samples taken at least 30 minutes apart)
* Were currently receiving treatment for hypogonadism in accordance with approved labelling, or in the Investigator's opinion are eligible to receive such treatment
* Body Mass Index (BMI) < 35.0 kg/m^2
* Haemoglobin levels at screening greater than or equal to 11.5 g/dL
* Adequate venous access on left or right arm to allow collection of a number of samples by venipuncture
* Ability to communicate with the trial staff, understand the Trial Information Sheet and sign the Written Informed Consent Forms; willing to follow the Protocol requirements and comply with Protocol restrictions and procedures

Exclusion Criteria:

* Current use of long acting testosterone injectables such as Nebido®
* Any significant history of allergy and/or sensitivity to the drug products or their excipients, including any history of sensitivity to testosterone and/or sunscreens
* Any clinically significant chronic illness or finding on screening physical exam and/or laboratory testing that makes it undesirable for the Investigator to enrol the trial subject in the trial and/or that in the Investigator's opinion, would interfere with the trial objectives or safety of the subject
* Chronic skin disorder (e.g. eczema, psoriasis) likely to interfere with transdermal drug absorption
* Men with suspected reversible hypogonadism
* Any man in whom testosterone therapy was contraindicated, which included those with:

  * Known or suspected carcinoma (or history of carcinoma) of the prostate or clinically significant symptoms of benign prostatic hyperplasia and/or clinically significant symptoms of lower urinary obstruction and International Prostate Symptom Scores (IPSS) scores of greater than or equal to 19
  * Known or suspected carcinoma (or history of carcinoma) of the breast
  * Severe liver disease (i.e. cirrhosis, hepatitis or liver tumours or liver function tests >2 times the upper limit of the normal range values)
  * Active deep vein thrombosis, thromboembolic disorders or a documented history of these conditions
  * Current significant cerebrovascular or coronary artery disease
  * Untreated sleep apnoea
  * Haematocrit of > 51
  * Untreated moderate to severe depression
* Men with clinically significant prostate exam (such as irregularities or nodules palpated) or clinically significant elevated serum Prostate Specific Antigen (PSA) levels (>4 ng/mL), or age adjusted reference range of PSA values
* Current or history of drug or alcohol abuse (more than 4 standard drinks per day and/or abnormal liver function tests >2 times the upper limit of the normal range values)
* Men taking concomitant medications (prescribed, over-the-counter or complementary) that would affect sex hormone binding globulin (SHBG) or testosterone concentrations or metabolism, warfarin, insulin, opiates, Gonadotropin-releasing hormone (GnRH), 5 alpha reductase inhibitors, propanolol, oxyphenbutazone, corticosteroids (except for physiological replacement doses), estradiol
* Men involved in sport in which there is screening for anabolic steroids
* Men with uncontrolled diabetes (haemoglobin A1c [HbA1c] greater than or equal to 10%)
* Men currently taking any investigational product, or have received an investigational product within 28 days prior to screening or 5 half-lives
* Any contraindication to blood sampling
* Subjects intending to have any surgical procedure during the course of the trial
* Subjects with a partner of child bearing potential who are not willing to use adequate contraception for the duration of the trial
* Subjects whose partners are pregnant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuscon, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shawnee Mission, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perth, Western Australia
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnsley
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle upon Tyne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swansea

REFERENCES:
- [Result] Wang C, Ilani N, Arver S, McLachlan RI, Soulis T, Watkinson A. Efficacy and safety of the 2% formulation of testosterone topical solution applied to the axillae in androgen-deficient men. Clin Endocrinol (Oxf). 2011 Dec;75(6):836-43. doi: 10.1111/j.1365-2265.2011.04152.x. PMID 21689131
- [Derived] Muram D, Ni X. Utility of a single serum testosterone measurement to determine response to topical testosterone replacement in hypogonadal men. Curr Med Res Opin. 2016;32(2):263-9. doi: 10.1185/03007995.2015.1117434. Epub 2015 Dec 15. PMID 26549704

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received Testosterone Metered Dose (MD)-Lotion for 120 days, at initial dose of 60 mg; may have had their dose adjusted up or down on Days 45 and 90 (3 were on 30mg; 97 on 60mg; 25 on 90mg; and 10 on 120mg). As primary outcome=subjects with normal testosterone at Day 120, results are presented for overall treatment group rather than dose.
Groups:
- Testosterone MD-Lotion: 30 mg to 120 mg of 2% Testosterone MD-Lotion administered topically once daily for 120 days.
Period: Overall Study
Arm/Group | Testosterone MD-Lotion
Started | 155
Completed | 135
Not Completed | 20
Not completed — Withdrawal by Subject | 9
Not completed — Non-Compliance of Study Drug | 3
Not completed — Lost to Follow-up | 2
Not completed — Non-Compliance with Site Directives | 1
Not completed — Sponsor Request | 1
Not completed — Screening Testosterone Levels >300 ng/dL | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 155
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 155
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Caucasian | 122
  African American | 6
  Hispanic | 13
  Other - Not Specified | 2
  Missing | 11
Region of Enrollment [Number; unit: participants]
  France | 11
  United States | 104
  Australia | 10
  Germany | 9
  United Kingdom | 10
  Sweden | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 29.53 (3.60)
Baseline Total Testosterone Level [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] | 196.73 (91.04)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 24-Hour Average Concentration [Cavg(0-24h)] Total Testosterone Within Normal Range at Day 120
Description: Cavg(0-24) is the average serum concentration calculated over the 24 hour period on Day 120. Calculated as the AUC(0-24) divided by 24 hours. Normal range for Total Testosterone was defined as 300 - 1050 nanograms per deciliter (ng/dL).
Time Frame: Day 120
Population: All participants who received at least one dose of study drug, had on-treatment data for at least one efficacy variable, and completed the Day 120 visit. Participants were also included if they withdrew prior to Day 120 because of adverse event or lack of efficacy (considered as treatment failures).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 138
percentage of participants | 84.1 [77.95 to 90.17]
Statistical Analysis 1: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.001, One-Sample Binomial (Wald) test, 2-sided

2. Secondary Outcome: Percentage of Participants With Maximum Serum Concentration (Cmax) >1500 ng/dL
Description: Cmax is the maximum observed serum concentration (>1500 ng/dL) during the 24 hour period on Day 120.
Time Frame: Day 120
Population: All participants who received at least one dose of study drug, had on-treatment data for at least one efficacy variable, and completed the Day 120 visit.
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 135
percentage of participants | 5.2

3. Secondary Outcome: Percentage of Participants With Cmax Between 1800 and 2500 ng/dL
Description: Cmax is the maximum observed serum concentration (between 1800 and 2500 ng/dL) during the 24 hour period on Day 120.
Time Frame: Day 120
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 135
percentage of participants | 3.0

4. Secondary Outcome: Percentage of Participants With Cmax >2500 ng/dL
Description: Cmax is the maximum observed serum concentration (>2500 ng/dL) during the 24 hour period on Day 120.
Time Frame: Day 120
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 135
percentage of participants | 0.7

5. Secondary Outcome: Percentage of Participants With Minimum Concentration (Cmin) <300 ng/dL
Description: Cmin is the minimum observed serum concentration (<300 ng/dL) during the 24 hour period on Day 120.
Time Frame: Day 120
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 135
percentage of participants | 64.4

6. Secondary Outcome: Change From Baseline to Endpoint in Psychosexual Daily Questionnaire
Description: Questions included: Sexual Desire (0=none to 7=very high), Overall Sexual Activity Score (calculated as average of weekly values on scale from 0=none to 7=Frequent), Erection Maintained for Satisfactory Duration (0=not satisfactory to 7=very satisfactory), and Positive and Negative Mood (individual mood variables on scale from 0=Not at all true to 7=very true). Positive mood: sum of 4 positive mood variables-alert, full of pep/energetic, friendly, and well/good (range from 0-28). Negative mood: sum of 5 negative mood variables-angry, irritable, sad/blue, tired, and nervous (range from 0-35).
Time Frame: Baseline, Day 120
Population: All participants who received at least one dose of study drug, had baseline and on-treatment data for at least one efficacy variable, and completed the Day 120 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 131
units on a scale
  Sexual Desire | 1.49 (1.84)
  Overall Sexual Activity Score | 0.94 (1.43)
  Erection Maintained for Satisfactory Duration | 1.11 (2.0)
  Positive Mood | 0.56 (1.25)
  Negative Mood | -0.50 (1.33)
Statistical Analysis 1: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is for Sexual Desire based on a two-sided, paired t-test comparing the Baseline and the Day 120 scores
Statistical Analysis 2: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is for Overall Sexual Activity Score based on a two-sided, paired t-test comparing the Baseline and the Day 120 scores
Statistical Analysis 3: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is for Erection Maintained for Satisfactory Duration based on a two-sided, paired t-test comparing the Baseline and the Day 120 scores
Statistical Analysis 4: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is for Positive Mood based on a two-sided, paired t-test comparing the Baseline and the Day 120 scores
Statistical Analysis 5: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value is for Negative Mood based on a two-sided, paired t-test comparing the Baseline and the Day 120 scores

7. Secondary Outcome: Change From Baseline to Endpoint in the 36-Item Short-Form Health Survey (SF-36)
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). MCS and PCS scores=0-100 (higher scores indicate better health status).
Time Frame: Baseline, Day 120
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 133
units on a scale
  Physical Component Score | 1.55 (7.72)
  Mental Component Score | 4.54 (9.20)
Statistical Analysis 1: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p = 0.0254, t-test, 2 sided — p-value for Physical Component Score based on a one-sample t-test comparing Day 120 and Baseline values
Statistical Analysis 2: Comparison: Testosterone MD-Lotion; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — p-value for Mental Component Score based on a one-sample t-test comparing Day 120 and Baseline values

8. Secondary Outcome: Change From Baseline to Endpoint in Fasting Insulin
Time Frame: Baseline, up to Day 120
Population: Participants enrolled in the study who had a baseline and a measurement at endpoint: Day 120, follow-up, or early withdrawal.
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 63
uIU/mL | 1.93 (12.02)

9. Secondary Outcome: Change From Baseline to Endpoint in Fasting Glucose
Time Frame: Baseline, up to Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 64
mg/dL | -0.41 (20.02)

10. Secondary Outcome: Change From Baseline to Endpoint in Prostate Specific Antigen (PSA)
Time Frame: Baseline, Day 120
Population: Participants enrolled in the study who had a baseline and a measurement at endpoint: Day 120.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 70
ng/mL | 0.13 (0.68)

11. Secondary Outcome: Change From Baseline to Endpoint in Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH)
Time Frame: Baseline, up to Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 54
mIU/mL
  Luteinizing Hormone (N=48) | -2.04 (5.36)
  Follicle Stimulating Hormone (N=54) | -2.41 (9.72)

12. Secondary Outcome: Change From Baseline to Endpoint in Estradiol
Time Frame: Baseline, up to Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 39
pg/mL | -2.16 (12.32)

13. Secondary Outcome: Change From Baseline to Endpoint in Haemoglobin
Time Frame: Baseline, up to Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 64
g/dL | 0.51 (1.08)

14. Secondary Outcome: Change From Baseline to Endpoint in Haematocrit
Description: Haematocrit: percentage of total blood volume made up of blood cells
Time Frame: Baseline, up to Day 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 64
percentage of red blood cells | 0.02 (0.04)

15. Secondary Outcome: Change From Baseline to Endpoint in Draize Score
Description: Draize score is a measurement of skin irritability of the application site based on erythema/eschar and oedema. Erythema/eschar scoring ranges from 0 (no erythema) to 4 (severe erythema [beet redness] to slight eschar formation [injuries in depth]). Oedema scoring ranges from 0 (no oedema) to 4 (severe oedema [raised more than 1 millimeter and extending beyond area of exposure]. The total Draize score ranges from 0 to 8.
Time Frame: Baseline, Day 120
Population: Participants enrolled in the study who had a baseline and a measurement at endpoint: Day 120.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone MD-Lotion
Number analyzed (Participants) | 135
units on a scale | 0 (0.17)

ADVERSE EVENTS:
Arm/Group | Testosterone MD-Lotion
Serious Adverse Events (participants affected / at risk) | 1/155
Other Adverse Events (participants affected / at risk) | 80/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone MD-Lotion (N=155)
Appendicitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone MD-Lotion (N=155)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Application site erythema (General disorders) | 8 (9)
Application site irritation (General disorders) | 11 (19)
Application site oedema (General disorders) | 2 (2)
Application site warmth (General disorders) | 2 (4)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Fungal infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (8)
Rhinitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Epicondylitis (Injury, poisoning and procedural complications) | 2 (2)
Blood glucose increased (Investigations) | 2 (2)
Haematocrit increased (Investigations) | 6 (6)
Haemoglobin increased (Investigations) | 2 (2)
Prostatic specific antigen increased (Investigations) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (11)
Migraine (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Anger (Psychiatric disorders) | 2 (4)
Anxiety (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Stress (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days